CLINICAL TRIAL: NCT03082703
Title: Impact of Text Messaging in the Management of Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashwani Singal,MD (Other)
Responsible Party: Sponsor-Investigator, Ashwani Singal,MD, PI, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X150420005
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: NAFLD and NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging (Experimental)
  Interventions: Behavioral: Text Messaging
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Text Messaging — Subjects contacted 3 times weekly via text messaging for the study period.
  Arms: Text Messaging

SUMMARY:
This randomized study aims at examining the impact of text messaging in the management of non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH), a disease frequently associated with obesity and varying components of metabolic syndrome including diabetes mellitus, hypertension, and dyslipidemia. With rising incidence of obesity in the US, NAFLD and NASH are rapidly increasing with currently the second etiology for liver transplantation in the US. The objectives of this protocol are to a) prospectively enroll patients with NAFLD and NASH; b) randomize them to receiving text messaging to help manage obesity and other components od metabolic syndrome in addition to standard clinical care or receiving only standard clinical care; and c) follow up these patients at the end of 3 months period for weight loss, blood pressure control, HBA1c, and liver enzymes. The immediate aim of this protocol is to develop the pilot data on the usefulness of text messaging in the management of NAFLD and NASH. The long-term goals of this research are to establish text messaging as a beneficial intervention in the management of weight loss and control of risk factors of NAFLD and improve outcomes of these patients with NAFLD and NASH.

DETAILED DESCRIPTION:
Patients will be recruited primarily from the outpatient Liver Kirklin Clinic setting.

1. Informed consent will be obtained by one of the investigators named in the protocol or by research coordinators involved with the study
2. Eligibility will be confirmed by interview and review of medical records using the inclusion and exclusion criteria as listed above.
3. Complete history and physical examination will be recorded especially for weight and body mass index, associated components of metabolic syndrome (diabetes, hypertension, and dyslipidemia), liver enzymes, and current medications list.
4. All procedures such as imaging, endoscopy, and liver biopsy will be done as part of standard routine care of these patients and no procedure will be done as part of this research study.
5. Patients would be randomized to standard clinical care or to text messaging in addition to standard clinical care. Standard clinical care includes obtaining data on history and physical examination, routine blood work as part of liver disease care, ultrasound and appropriate any other liver imaging as needed for patient care, counseling for at least 7-10% weight loss with discussion on strategies to achieve this, management of other risk factors including diabetes, hypertension, and dyslipidemia, and counseling for compliance to taking medications and following up on future clinic visits. The study investigator would be blinded to the randomization and which group the patient is randomized to.
6. Patients would be followed at the end of 6 months period for assessing the study outcomes as detailed earlier. Follow up for patients with stable liver disease is usually done every 3-6 months. No additional clinic visits would be needed for this study.
7. During these 6 months, patients would receive standard text messages as detailed later. Patients will use their own cell phone to receive the text messages and reply to these messages. There will be no additional intervention or device needed for this study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of NAFLD or NASH as determined with presence of steatosis and/or elevated liver enzymes, exclusion of other causes of liver disease, and history of alcohol use less than 10 g/d.
2. Age >18 years
3. Established patient at the UAB Kirklin clinic for at least 3-6 months
4. Ownership of cell phone with text messaging service
5. Ability to read and send text message

Exclusion Criteria:

1. Failure to meet the inclusion criteria.
2. Any medical, psychiatric, or social conditions that, in the opinion of the investigators, would make participation in this protocol not in the best interest of the subject
3. Refusal to consent for the study
4. Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 months

IPD SHARING:
Plan to Share IPD: No